CLINICAL TRIAL: NCT06788951
Title: Investigation of the Effects of Oral Carbohydrate Solution Given to Patients Before Coronary Artery Bypass Graft Surgery on Postoperative Nausea and Vomiting, Feeling of Hunger and Thirst, Physiological Parameters and Recovery
Brief Title: The Effect of Oral Carbohydrate Inhalation Given to Patients Before Coronary Artery Bypass Graft Operation on Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Bozkurt (Other)
Responsible Party: Sponsor-Investigator, Yasemin Bozkurt, Nurse, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Ybozkurt
Record Dates: First submitted 2024-12-27; First posted 2025-01-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Surgery
Keywords: Surgery; ERAS; Nursing; Cardiovascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral carbohydrate solution was administered preoperatively (Experimental): The experimental group will be given 800 ml of ora carbohydrate solution until midnight before surgery and 400 ml 2 hours before surgery. Patient Information Form will be collected from the patients before surgery. After the surgery, the Visual Comparison Scale, Physiological Parameters and Blood Glucose Monitoring, Form Postoperative Recovery Index (Turkish Version), and the Number and Dosage of Antiemetic Drugs Taken in the Postoperative 24 Hours form will be used.
  Interventions: Dietary Supplement: administration of oral carbohydrate solution to patients before coronary artery bypass graft surgery
- Flavored Water Applied Before Surgery (Placebo Comparator): The placebo group will receive 800 ml of flavored water until midnight before surgery and 400 ml 2 hours before surgery. A Patient Information Form will be collected from the patients before surgery. After the surgery, the Visual Comparison Scale, Physiological Parameters and Blood Glucose Monitoring Form, Postoperative Recovery Index (Turkish Version) and the Number and Dosage of Antiemetic Drugs Taken in 24 Hours Postoperatively will be used.
  Interventions: Other: giving flavored water to patients before coronary artery bypass graft surgery
- No Preoperative Intervention (No Intervention): No intervention will be made to patients who will undergo surgery. Patient Information Form will be collected from the patients before surgery. After the surgery, the Visual Comparison Scale, Physiological Parameters and Blood Glucose Monitoring Form, Postoperative Recovery Index (Turkish Version) and the Number and Dosage of Antiemetic Drugs Taken in 24 Hours Postoperatively will be used.

INTERVENTIONS:
Dietary Supplement: administration of oral carbohydrate solution to patients before coronary artery bypass graft surgery — Oral carbohydrate solution will be administered to patients before coronary artery bypass graft operation and its effects on postoperative nausea-vomiting, hunger, thirst, physiological parameters and recovery will be evaluated.
  Arms: Oral carbohydrate solution was administered preoperatively
Other: giving flavored water to patients before coronary artery bypass graft surgery — The effects of flavored water given to patients before coronary artery bypass graft operation on postoperative nausea-vomiting, hunger and thirst,
  Arms: Flavored Water Applied Before Surgery

SUMMARY:
The aim of this study was to investigate the effect of oral carbohydrate solution given to patients before coronary artery bypass graft surgery on nausea-vomiting, hunger, thirst, physiologic parameters and recovery.

The study will be completed with a total of 120 participants, 40 control, 40 placebo and 40 experimental.

As a randomization method, simple randomization method will be used to provide an equal number of samples in three groups and patients will be informed verbally about the study and written informed consent will be obtained from patients who agree.

In this study, the effects of oral carbohydrate solution administration on nausea and vomiting, hunger, thirst, physiologic parameters and recovery were evaluated before coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Experimental: Oral administration of carbohydrate solution Patients will receive 800 ml of oral carbohydrate solution until midnight before surgery and 400 ml until 2 hours before surgery. Patients will be administered a Patient Information Form before surgery. Postoperative Recovery Index (Turkish Version), Visual Comparison Scale, Physiologic Parameters and Blood Glucose Monitoring Form and Number and Dosage of Antiemetic Drugs Taken in 24 Hours Postoperatively will be applied.

Placebo: Administration of flavored water Patients will be given 800 ml of flavored water until midnight before surgery and 400 ml of flavored water until 2 hours before surgery. Patients will be given a Patient Information Form before surgery. Postoperative Recovery Index (Turkish Version), Visual Comparison Scale, Physiologic Parameters and Blood Glucose Monitoring Form and Number and Dosage of Antiemetic Drugs Taken in 24 Hours Postoperatively will be applied.

Control: No intervention Patients will be administered a Patient Information Form before surgery. Postoperative Recovery Index (Turkish Version), Visual Comparison Scale, Physiologic Parameters and Blood Glucose Monitoring Form and Number and Dosage of Antiemetic Drugs Taken in 24 Hours Postoperatively will be applied.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Planned coronary artery bypass graft surgery
* Volunteering to participate in the research

Exclusion Criteria:

* Under 18 years of age
* Not planned coronary artery bypass graft surgery
* Not volunteering to participate in the research
* Cases received as an emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | Up to 24 weeks
  The personal information form used in the data collection process consists of demographic characteristics of the individuals such as age, gender, marital status, occupation, educational status and employment status, as well as health-related conditions of the patients such as chronic diseases and past surgical history.

SECONDARY OUTCOMES:
Postoperative Recovery Index (Turkish Version) | Up to 24 weeks
  The Postoperative Recovery Index (PRAI) used in the validity and reliability study conducted by Butler et al. (2012) consists of 25 items. This index includes psychological symptoms, physical activities, general symptoms, bowel symptoms and craving symptoms. In scoring the questionnaire, the scores of the items in each subscale are summed and a subscale score is obtained by taking the arithmetic mean. The ASI overall questionnaire score is calculated by taking the arithmetic mean of the total score over 25 items. Higher scores on the index indicate that postoperative recovery is more difficult and lower scores indicate that recovery is easier. The minimum score value in each parameter of this scale is 0 and the maximum score value is 5. In this study, the Cronbach's alpha coefficient of the ASIQ was 0.97, 0.90 for the psychological symptoms subscale, 0.83 for the physical activity subscale and 0.98 for the discomfort subscale.

OTHER OUTCOMES:
Visual Benchmark Scale | Up to 24 weeks
  This scale is used to measure various parameters such as hunger, thirst, nausea and vomiting. The scale value ranges from 0 to 10, with an increase in value indicating an increase in the relevant parameters. The minimum score on this scale is 0 and the maximum score is 10.
Number and Dosage of Antiemetic Drugs Taken in 24 Hours Postoperatively | Up to 24 weeks
  This questionnaire was used to assess the dose and number of antiemetic drugs used in the postoperative period. This questionnaire was used to measure patients' nausea and vomiting in the postoperative period. Scoring was evaluated on a scale of 0-10. The closer the score range was to 10, the higher the discomfort rate of the patients, while a score range closer to 0 indicated less discomfort.
Physiological Parameters and Blood Glucose Monitoring Form | Up to 24 weeks
  This form is a comprehensive tracking tool for monitoring patients' vital signs. It includes regular recording of important parameters such as blood pressure, pulse rate, respiratory rate, oxygen saturation, body temperature and blood sugar. These regular measurements allow monitoring changes in the surgical process and the recovery process. The optimal value range of blood pressure is 120/80 mg/dl, pulse rate range is between 60-100 per minute, respiratory rate optimal value is between 12-20 per second, oxygen saturation optimal value is between 95-100, body temperature value is between 36-37'C, and blood glucose value is close to 90-140 values are close to the optimal value and the effect of oral carbohydrate solution on postoperative physiological parameters is positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin BOZKURT, Van, Tuşba, Turkey (Türkiye)